CLINICAL TRIAL: NCT02069912
Title: Multifaceted Depression and Cardiovascular Program for Low-Income Patients
Brief Title: Multifaceted Depression and Cardiovascular Program
Acronym: MDCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Los Angeles County Department of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: USCIRB-HS-06-00420; CA Health Care Foundation (Other Grant/Funding Number: California Health Care Foundation)
Record Dates: First submitted 2014-02-20; First posted 2014-02-24 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2014-02

CONDITIONS: Depression; Depressive Disorder; Behavioral Symptoms; Mood Disorders
Keywords: Major Depression; Heart Disease; Hispanics; Collaborative Depression Care Management
MeSH Terms: conditions — Depression; Depressive Disorder; Behavioral Symptoms; Mood Disorders; Depressive Disorder, Major; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Collaborative depression care (Experimental): All enrolled patients will receive collaborative depression care management.
  Interventions: Behavioral: Collaborative depression care management

INTERVENTIONS:
Behavioral: Collaborative depression care management — Collaborative depression care management will include acute depression treatment with antidepressant medication and/or counseling sessions based on structured problem solving therapy. Participants will also receive supportive patient navigation services and maintenance/relapse telephone monitoring. Counseling treatment will include 8 weekly 45-minute counseling sessions that are culturally and health literacy adapted for the study population. The length of medication treatment will depend upon participants' severity of depression and may last up to 12 months.

SUMMARY:
1. Implement an evidence-based structured care approach that includes screening; acute treatment and relapse prevention follow-up tailored for public sector clinics and low-income and minority patients.
2. Adapt an evidence-based collaborative care model for primary care, implement the adapted model, evaluate and further refine the model based on the pilot experience, and produce and disseminate a detailed manual for use in public sector clinics.
3. Evaluate Multifaceted Depression and Cardiovascular Program (MDCP) in an open trial to determine: its acceptance by patients, medical providers, and organizational decision-makers; patient depression treatment adherence; its direct cost; and the size and variability of change from baseline in the primary outcome measures: depressive symptoms, functional status, quality of life, health service use, and cardiac status at 6 and 12 month follow-up.

DETAILED DESCRIPTION:
The pilot open trial was conducted to evaluate the effectiveness of a health services quality improvement intervention, Multifaceted Depression and Cardiovascular Program (MDCP), on reduction of major depressive disorder, adherence to recommended cardiac exercise and diet self-care regimens and appointment keeping, blood pressure and low density lipid levels, functional status, quality of life and use of health services among low-income, predominantly Hispanic adults with congestive heart failure (CHF) or other cardiac disease such as coronary artery disease (CAD) in public sector community-based primary care clinics. The study was based on key observations from recent studies: 1) Patients with cardiac conditions are more likely to experience clinically significant depressive symptoms than the general population, with depression being associated with poor cardiac outcomes; 2) depression rates are high among Hispanics with chronic illness; 3) Minority patients are less likely to receive care for depression, but benefit with culturally appropriate care enhancements; and 4) depression co-morbid with cardiac conditions is likely to be persistent. Low-income patient needs, depression illness characteristics, and public care system resources call for a multifaceted, collaborative chronic disease management model of depression care. MDCP is aimed at positively affecting depression and cardiac outcomes by reducing known patient, provider, and system barriers to care.

Participation in this study will last 12 months. All participants will first undergo baseline assessments that will include a 40-minute interview about personal health and feelings. All study participants will receive collaborative depression care management. They will first be provided with information about depression treatment. Participants will then have the option of choosing between two depression treatments: counseling or antidepressant medications. Participants who choose to receive treatment with counseling will receive eight weekly 45-minute counseling sessions, conducted either on the phone or at the clinic. During these sessions, participants will undergo structured problem solving therapy (PST) and will learn strategies to manage their depressive symptoms. Participants who choose to receive treatment with antidepressant medication will be prescribed medication by a study doctor and will be monitored for any side effects throughout treatment. Medication treatment may last up to 12 months but will depend upon participants' severity of depression. After completing medication treatment, participants will be offered PST counseling. All study participants will also receive supportive patient navigation services and maintenance/relapse telephone monitoring.

All participants will undergo follow-up phone interviews about their status at months 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for clinically significant depression based on a score of ≥ 2 for one of the two cardinal depression symptoms (depressed mood or loss of interest) and a Patient Health Questionnaire-9 total score of ≥ 10
* Patient with heart disease
* Has attended Los Angeles County Department of Health Services Comprehensive Health Clinics or the Cardiology Clinic at Los Angeles County+University of Southern California Medical Center

Exclusion Criteria:

* Current suicidal ideation
* Score of 8 or greater on the Alcohol Use Disorders Identification Test (AUDIT)
* Recent use of lithium or antipsychotic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2006-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms reduction | Measured at months 6 and 12
  Achieve minimum a 50% reduction in depressive symptoms from baseline at 6- and 12-month follow-up

SECONDARY OUTCOMES:
Improvement in quality of life | Measured at months 6 and 12
  Change score in quality-of-life 12-item Short-Form Health Survey, Minnesota Living with Heart Failure, Sheehan Disability Scale outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen R Ell, DSW, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California School of Social Work, Los Angeles, California, United States

REFERENCES:
- [Derived] Ell K, Oh H, Lee PJ, Guterman J. Collaborative health literate depression care among predominantly Hispanic patients with coronary heart disease in safety net care. Psychosomatics. 2014 Nov-Dec;55(6):555-65. doi: 10.1016/j.psym.2014.03.007. Epub 2014 Mar 26. PMID 25262042